CLINICAL TRIAL: NCT03379753
Title: The Influence of Postoperative Environment on Patient Satisfaction and Perception of Care Following Pelvic Reconstructive Surgery
Brief Title: Postoperative Environment on Pain Following Pelvic Reconstructive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-076
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Those patients randomized to intervention group will be exposed to the diad of music and positive images in a private hospital room in addition to receiving standard care.
  Interventions: Other: music and positive images
- Control group (No Intervention): Those patients randomized to control group will receiving standard care in a private hospital room with an un-modified post operative environment.

INTERVENTIONS:
Other: music and positive images — The diad of misic and positive image will be administered to the standard care by adding a Bluetooth capable speaker with selections of music and a soothing nature landscape into the hospital room.
  Arms: Intervention group

SUMMARY:
This study is to determine if patients following prolapse repair including vaginal vault suspension have decreased pain measured via a visual analog scale (VAS) on postoperative day one and just prior to discharge when exposed to the diad of music and positive images compared to patients receiving standard care.

DETAILED DESCRIPTION:
Over the past decade, interest has grown in improving the patient experience. As part of this movement, studies have sought to evaluate the mechanisms by which the postoperative environment affects a patient's outcome and perception of healing.

Literature review reveals efforts by both medical and design teams towards improving the experience of the patient and developing an environment that promotes healing. Changes to the physical environment have been shown to have an impact on satisfaction. These parameters have included music and art. Considering the effort that is now going into improving the patient experience and developing this theory of healing spaces, there has yet to be a randomized controlled trial evaluating these alternative therapies in the urogynecologic patient population. Although each of these modalities appears beneficial, we believe that a combination of these would be even more useful. Indeed, these treatments are also relatively easy to implement without undue cost or burden to the hospital. This study seeks to determine the influence of applying music and art to the post operative environment for patients recovering from major urogynecologic surgery on pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-85 years of age
* English speaking
* Undergoing surgery for pelvic organ prolapse to include an apical vaginal vault suspension by a physician at Cincinnati Urogynecology Associates, TriHealth
* Concomitant procedures such as hysterectomy, suburethral sling, anterior or posterior colporrhaphy, bilateral salpingectomy or salpingooophorectomy will be included
* Ability to complete the questionnaires and provide consent
* Willingness to listen to music at the minimum recommended time intervals

Exclusion Criteria:

* Unwillingness to participate in the study
* Physical or mental impairment that would affect the subject's ability to utilize the modified environment such as deafness, blindness or dementia
* Patients who take daily narcotics or NSAIDS
* Patients with history of Drug or Alcohol Abuse
* Patients with chronic pain syndromes
* Non English speaking
* Patients that do not undergo a vaginal apical suspension procedure

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 61 | 71
Completed | 46 | 46
Not Completed | 15 | 25
Not completed — Withdrawal by Subject | 2 | 1
Not completed — not having correct procedure | 1 | 2
Not completed — No primary outcome | 12 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.4) | 63.6 (9.6) | 63.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 92
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 44 | 43 | 87
  Black/African American | 1 | 2 | 3
  Hispanic | 0 | 1 | 1
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Score for Pain
Description: VAS score for pain administered following breakfast on post-operative day one. The VAS was100 millimeter (mm) scale with 'no pain' on the far left represented as 0 mm and 'most pain' on the far right equating to 100 mm.
Time Frame: following breakfast on Post-operative day one
Measure: Median (Full Range); unit: millimeter (mm)
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 46 | 46
millimeter (mm) | 28.0 [0 to 86] | 24.5 [0 to 81]
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Other; p = 0.57, Wilcoxon (Mann-Whitney); U statistic = 984.5

ADVERSE EVENTS:
Time Frame: 2 week post-op
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT03379753/Prot_SAP_000.pdf